CLINICAL TRIAL: NCT02622607
Title: Preventive Effects of Zoledronic Acid on Bone Metastasis in Patients With Stage IIIB and IV Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZOL
Record Dates: First submitted 2015-11-30; First posted 2015-12-04 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Lung Cancer
Keywords: ZOL; Prevention; lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ZOL (Experimental): Zoledronic acid 4 mg intravenous infusion over at least 15 minutes every 3 months for 12 months.
  Interventions: Drug: Zoledronic acid
- Control (No Intervention): No investigational treatment

INTERVENTIONS:
Drug: Zoledronic acid — Zoledronic acid 4 mg in 5 mL concentrated solution prepared with 100 mL calcium free infusion solution (0.9 % sodium chloride)
  Other Names: Zometa
  Arms: ZOL

SUMMARY:
Bone metastases are common in patients with advanced lung cancer and can have devastating consequences. Preventing or delaying bone metastases may improve outcomes. Bisphosphonates are inhibitors of osteoclast-mediated bone resorption. The current indications for bisphosphonates include the treatment of metabolic disorders of bone metabolism (e.g., osteoporosis and Paget's disease), the treatment of hypercalcaemia of malignancy (HCM), and the prevention of skeletal-related events(SREs）from malignant bone disease. Clinical trials also confirm that bisphosphonates, and zoledronic acid（ZOL) in particular, can prevent bone loss from cancer treatment.There is also emerging evidence that the benefits of bisphosphonate therapy in the oncology setting are more extensive. This study will evaluate whether the addition of ZOL 4 mg every 3 months for up to 1 years in patients with stage IIIB/IV lung cancer could reduce the rate of bone metastases ,improve progression-free survival (PFS) and overall survival(OS), and delay time to bone metastases .

DETAILED DESCRIPTION:
Bone metastases are common in patients with advanced lung cancer and can have devastating consequences. which can lead to pain, decreased mobility and skeletal complications .Preventing or delaying bone metastases may improve outcomes. Bisphosphonates are inhibitors of osteoclast-mediated bone resorption. The current indications for bisphosphonates include the treatment of metabolic disorders of bone metabolism (e.g., osteoporosis and Paget's disease), the treatment of hypercalcaemia of malignancy (HCM), and the prevention of SREs from malignant bone disease. Clinical trials also confirm that bisphosphonates, and zoledronic acid in particular, can prevent bone loss from cancer treatment.There is also emerging evidence that the benefits of bisphosphonate therapy in the oncology setting are more extensive. This study will evaluate whether the addition of ZOL 4 mg every 3 months for up to 1 years in patients with stage IIIB/IV lung cancer could reduce the rate of bone metastases ,improve progression-free survival (PFS) and overall survival(OS), and delay time to bone metastases .

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70 years of age, male or female
2. histologically or cytologically confirmed stage IIIB or IV lung cancer at diagnosis
3. no evidence of bone metastatic lesions was radiographically confirmed by bone scintigraphy
4. life expectancy of ≥6 months
5. adequate renal, hematologic, and hepatic
6. Eastern Cooperative Oncology Group(ECOG) performance status≤2
7. All patients provided written informed consent

Exclusion Criteria:

1. Treatment with other bisphosphonates
2. Presence of brain metastases
3. Be allergic to ZOL
4. attending other unlisted drug clinical trials,currently.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-01; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Bone Metastases at 12 Months | Months 12
  Percentage of participants developing at least 1 bone metastasis, whether or not symptomatic. Bone scans were scheduled at screening and at 6-monthly intervals after study entry, or when symptoms suggested the presence of bone metastases. Positive bone scans required confirmation by x-ray, magnetic resonance imaging (MRI), or computed tomography (CT).

SECONDARY OUTCOMES:
Progression-Free Survival | Up to 24 months
  Progression-free survival is defined as the time from randomization to the date of the first documented progression or recurrence of disease or death from any cause. Time to disease progression (TTP) was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) guidelines with evaluations every 3 months.
Percentage of Participants With Overall Survival | Months 6, 12, 18, and 24 ]

CONTACTS AND LOCATIONS:
Overall Officials: He-Long Zhang, M.D., Study Chair — Department of Oncology，Tangdu Hospital
Locations (1):
- Department of Oncology，Tangdu Hospital，Fourth Millitary Medical University, Xi'an, Shaanxi, China